CLINICAL TRIAL: NCT00262119
Title: MINERVA: MINimizE Right Ventricular Pacing to Prevent Atrial Fibrillation and Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MNV-20-171005
Record Dates: First submitted 2005-12-04; First posted 2005-12-06 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2016-03

CONDITIONS: Atrial Fibrillation; Heart Failure, Congestive
Keywords: Physiological pacing; Antitachycardia pacing therapies
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Control Group (Active Comparator): PM programming according to actual clinical practice
  Interventions: Device: Pacemaker Medtronic EnRhythm
- MVP Only (Active Comparator): PM programming according to actual clinical practice + MVP algorithm ON
  Interventions: Device: Pacemaker Medtronic EnRhythm
- DDDRP (Active Comparator): PM programming according to actual clinical practice + MVP algorithm ON + Atrial fibrillation therapies ON
  Interventions: Device: Pacemaker Medtronic EnRhythm

INTERVENTIONS:
Device: Pacemaker Medtronic EnRhythm — Pacemaker specific programming

SUMMARY:
The aim of this study is to test the impact of the managed ventricular pacing (MVP) mode and atrial preventive and antitachycardia pacing therapies on the reduction of a composite clinical outcome composed of any death, permanent atrial fibrillation, and cardiovascular hospitalizations.

DETAILED DESCRIPTION:
Kristensen et al. reported that AAIR pacing reduces atrial fibrillation (AF) development compared to DDDR pacing in sinus node disfunction patients.

Several authors have shown that, in patients with intact AV conduction, unnecessary chronic RV pacing can cause detrimental effects such as AF, left ventricular (LV) dysfunction and congestive heart failure. These findings arose the hypothesis that the non-physiologic nature of ventricular pacing may result in electrophysiological and LV remodeling changes that have potentially deleterious long-term effects.

The MVP mode, present in the Medtronic pacemaker EnRhythm, provides atrial based pacing with ventricular backup. It operates in true AAI(R) mode, it provides ventricular backup in case of a single conduction loss and converts to DDD(R) mode in case of persistent loss of AV conduction.

Aim of this study is to test the impact of the MVP pacing mode and atrial preventive and antitachycardia pacing therapies on the reduction of a composite clinical outcome composed by any death, permanent AF, cardiovascular hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Class I/Class II indications for dual chamber pacing
* Previous implant of an EnRhythm dual chamber implantable pulse generator (IPG) since maximum 2 weeks
* History of atrial arrhythmias (at least one electrocardiogram [ECG] or Holter documented episodes in the last 12 months)

Exclusion Criteria:

* Less than 18 years of age
* Pregnancy
* Unwilling or unable to give informed consent or to commit to follow-up schedule
* Medical conditions that preclude protocol required testing or limit study participation
* Enrolled or intend to participate in another clinical trial during the course of this study
* A life expectancy of less than 2 years
* Patient is a candidate for an implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy (CRT) device implant
* Anticipated major cardiac surgery within the course of this study
* Permanent III degree AV-block or history of AV node ablation
* History of permanent AF (as defined below)
* AF ablation (left pulmonary veins) or other cardiac surgery < 3 months
* Prior implant of defibrillator device or pacemaker (apart from EnRhythm IPG implanted within two weeks)
* Uncontrolled hyperthyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2006-02; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Padeletti, Prof., Principal Investigator — Ospedale Careggi - Firenze; Giuseppe Boriani, Dr., Principal Investigator — Ospedale Sant'Orsola - Bologna; Luis Mont, Dr., Principal Investigator — Hospital Clinic of Barcelona; Reinhard C Funck, Dr., Principal Investigator — Philipps University Hospital - Marburg; Carsten W Israel, Dr., Principal Investigator — J. W. Goethe University Hospital - Frankfurt; Helmut Pürerfellner, Dr., Principal Investigator — Elisabethinen Hospital; Antonis S Manolis, Prof., Principal Investigator — Evagelismos Hospital - Athens; André Pisapia, Dr, Principal Investigator — Hôpital Saint-Joseph - Marseille; Raymond Tukkie, Dr, Principal Investigator — Kennemer Gasthuis
Locations (1):
- Medtronic Italia S.p.A., Rome, Italy

REFERENCES:
- [Background] Connolly SJ, Kerr CR, Gent M, Roberts RS, Yusuf S, Gillis AM, Sami MH, Talajic M, Tang AS, Klein GJ, Lau C, Newman DM. Effects of physiologic pacing versus ventricular pacing on the risk of stroke and death due to cardiovascular causes. Canadian Trial of Physiologic Pacing Investigators. N Engl J Med. 2000 May 11;342(19):1385-91. doi: 10.1056/NEJM200005113421902. PMID 10805823
- [Background] Lamas GA, Lee KL, Sweeney MO, Silverman R, Leon A, Yee R, Marinchak RA, Flaker G, Schron E, Orav EJ, Hellkamp AS, Greer S, McAnulty J, Ellenbogen K, Ehlert F, Freedman RA, Estes NA 3rd, Greenspon A, Goldman L; Mode Selection Trial in Sinus-Node Dysfunction. Ventricular pacing or dual-chamber pacing for sinus-node dysfunction. N Engl J Med. 2002 Jun 13;346(24):1854-62. doi: 10.1056/NEJMoa013040. PMID 12063369
- [Background] Mattioli AV, Vivoli D, Mattioli G. Influence of pacing modalities on the incidence of atrial fibrillation in patients without prior atrial fibrillation. A prospective study. Eur Heart J. 1998 Feb;19(2):282-6. doi: 10.1053/euhj.1997.0616. PMID 9519322
- [Background] Andersen HR, Nielsen JC, Thomsen PE, Thuesen L, Mortensen PT, Vesterlund T, Pedersen AK. Long-term follow-up of patients from a randomised trial of atrial versus ventricular pacing for sick-sinus syndrome. Lancet. 1997 Oct 25;350(9086):1210-6. doi: 10.1016/S0140-6736(97)03425-9. PMID 9652562
- [Background] Kristensen L, Nielsen JC, Mortensen PT, Pedersen OL, Pedersen AK, Andersen HR. Incidence of atrial fibrillation and thromboembolism in a randomised trial of atrial versus dual chamber pacing in 177 patients with sick sinus syndrome. Heart. 2004 Jun;90(6):661-6. doi: 10.1136/hrt.2003.016063. PMID 15145874
- [Background] Nielsen JC, Andersen HR, Thomsen PE, Thuesen L, Mortensen PT, Vesterlund T, Pedersen AK. Heart failure and echocardiographic changes during long-term follow-up of patients with sick sinus syndrome randomized to single-chamber atrial or ventricular pacing. Circulation. 1998 Mar 17;97(10):987-95. doi: 10.1161/01.cir.97.10.987. PMID 9529267
- [Background] Nielsen JC, Kristensen L, Andersen HR, Mortensen PT, Pedersen OL, Pedersen AK. A randomized comparison of atrial and dual-chamber pacing in 177 consecutive patients with sick sinus syndrome: echocardiographic and clinical outcome. J Am Coll Cardiol. 2003 Aug 20;42(4):614-23. doi: 10.1016/s0735-1097(03)00757-5. PMID 12932590
- [Derived] Boriani G, Tukkie R, Manolis AS, Mont L, Purerfellner H, Santini M, Inama G, Serra P, de Sousa J, Botto GL, Mangoni L, Grammatico A, Padeletti L; MINERVA Investigators. Atrial antitachycardia pacing and managed ventricular pacing in bradycardia patients with paroxysmal or persistent atrial tachyarrhythmias: the MINERVA randomized multicentre international trial. Eur Heart J. 2014 Sep 14;35(35):2352-62. doi: 10.1093/eurheartj/ehu165. Epub 2014 Apr 25. PMID 24771721
- [Derived] Funck RC, Boriani G, Manolis AS, Puererfellner H, Mont L, Tukkie R, Pisapia A, Israel CW, Grovale N, Grammatico A, Padeletti L; MINERVA Study Group. The MINERVA study design and rationale: a controlled randomized trial to assess the clinical benefit of minimizing ventricular pacing in pacemaker patients with atrial tachyarrhythmias. Am Heart J. 2008 Sep;156(3):445-51. doi: 10.1016/j.ahj.2008.05.004. PMID 18760124

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was between February 2006 and April 2010. Patients were enrolled in cardiology departments.
Pre-assignment Details: A total of 1300 patients were enrolled in the study. Enrollment was followed by a 1-month run-in period. Patients with ventricular pacing ≥ 95% on device check in the run-in period were excluded from the study. At the end of the run-in period, randomization was performed. In all, 1166 patients were randomized and followed up.
Period: Overall Study
Arm/Group | Control Group | MVP Only | DDDRP
Started | 385 | 398 | 383
Completed | 327 | 328 | 325
Not Completed | 58 | 70 | 58
Not completed — Lost to Follow-up | 38 | 51 | 42
Not completed — Death | 20 | 19 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | MVP Only | DDDRP | Total
Number analyzed (Participants) | 385 | 398 | 383 | 1166
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (9) | 74 (9) | 74 (9) | 74 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 188 | 210 | 578
  Male | 205 | 210 | 173 | 588
Region of Enrollment [Number; unit: participants]
  Italy | 203 | 211 | 202 | 616
  Netherlands | 41 | 43 | 39 | 123
  Spain | 16 | 18 | 17 | 51
  Portugal | 43 | 44 | 44 | 131
  Austria | 15 | 14 | 15 | 44
  France | 0 | 1 | 1 | 2
  Germany | 8 | 5 | 3 | 16
  Greece | 23 | 25 | 25 | 73
  Hong Kong | 1 | 1 | 1 | 3
  Israel | 7 | 7 | 8 | 22
  Kuwait | 2 | 4 | 3 | 9
  Russian Federation | 10 | 11 | 9 | 30
  Slovakia | 5 | 5 | 6 | 16
  Switzerland | 9 | 7 | 7 | 23
  Taiwan | 2 | 2 | 3 | 7

OUTCOME MEASURES:

1. Secondary Outcome: Death for All Causes at 2 Years
Description: Incidence, estimated via Kaplan Meier survival analysis, of death for any cause at 2 years
Time Frame: 2 years
Population: The analysis was intention to treat therefore all randomized patients were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Control Group | MVP Only | DDDRP
Number analyzed (Participants) | 383 | 398 | 383
percentage of participants | 5.6 [3.6 to 8.5] | 5.1 [3.3 to 7.9] | 4.6 [2.8 to 7.3]

2. Secondary Outcome: Incidence of Permanent Atrial Fibrillation at 2 Years
Description: Incidence, estimated via Kaplan Meier survival analysis, of permanent atrial fibrillation at 2 years
Time Frame: 2 years
Population: The analysis was intention to treat therefore all randomized patients were analysed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Control Group | MVP Only | DDDRP
Number analyzed (Participants) | 383 | 398 | 385
percentage of participants | 9.2 [6.6 to 12.7] | 7.7 [5.3 to 11.0] | 3.8 [2.2 to 6.5]

3. Secondary Outcome: Incidence of Cardiovascular Hospitalizations at 2 Years
Description: Incidence, estimated via Kaplan Meier survival analysis, of cardiovascular hospitalizations at 2 years
Time Frame: 2 years
Population: Analysis was intention to treat therefore all randomized patients were analysed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Control Group | MVP Only | DDDRP
Number analyzed (Participants) | 383 | 398 | 385
percentage of participants | 16.8 [13.3 to 21.2] | 13.7 [10.5 to 17.7] | 15.2 [11.8 to 19.4]

4. Secondary Outcome: Burden of Composite Clinical Endpoint
Time Frame: 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Subjects' Symptoms
Time Frame: 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Heart Failure Medications
Time Frame: 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Cumulative Percentage of Ventricular Pacing
Time Frame: 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Cardiovascular Death
Time Frame: 2 years
Reporting Status: Not Posted

9. Secondary Outcome: Any Hospitalization
Time Frame: 2 years
Reporting Status: Not Posted

10. Secondary Outcome: Atrial Fibrillation Burden
Time Frame: 2 years
Reporting Status: Not Posted

11. Secondary Outcome: Persistent Atrial Fibrillation (AF)
Time Frame: 2 years
Reporting Status: Not Posted

12. Secondary Outcome: Adverse Events
Time Frame: 2 years
Reporting Status: Not Posted

13. Secondary Outcome: Development of Atrioventricular (AV) Block and Pacemaker Dependency
Time Frame: 2 years
Reporting Status: Not Posted

14. Secondary Outcome: Predictors of Stroke, Transient Ischemic Attack (TIA) and Arterial Embolism
Time Frame: 2 years
Reporting Status: Not Posted

15. Secondary Outcome: Echocardiogram Data About Left Ventricular Fractional Shortening and Ejection Fraction and Left Atrium Dilatation
Time Frame: 2 years
Reporting Status: Not Posted

16. Secondary Outcome: Clinical Outcome in All the Patients With MVP ON Between Patients With Optimized AV-delay and Patients Without Optimized AV-delay
Time Frame: 2 years
Reporting Status: Not Posted

17. Secondary Outcome: Time to Development of the Composite Endpoint Between All Randomized Subjects in the Three Arms in Subgroups of Patients
Time Frame: 2 years
Reporting Status: Not Posted

18. Secondary Outcome: Frequency, Type, and Associated Cost of Health Care Utilization and Utility
Time Frame: 2 years
Reporting Status: Not Posted

19. Primary Outcome: Composite Endpoint Composed by Death for Any Cause, Cardiovascular Hospitalization or Permanent AF at 2 Years
Description: The outcome measurement is the 2 years incidence, calculated by Kaplan Meier survival analysis, of the composite endpoint composed by death for any cause, cardiovascular hospitalization or permanent AF.
Time Frame: 2 years
Population: Analysis was intention to treat therefore all randomized patients were considered in the analyses
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Control Group | MVP Only | DDDRP
Number analyzed (Participants) | 385 | 398 | 383
percentage of participants | 28.0 [23.7 to 32.9] | 23.1 [19.1 to 27.8] | 21.5 [17.6 to 26.2]

ADVERSE EVENTS:
Arm/Group | Control Group | MVP Only | DDDRP
Serious Adverse Events (participants affected / at risk) | 180/385 | 165/398 | 169/383
Other Adverse Events (participants affected / at risk) | 0/385 | 0/398 | 0/383
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=385) | MVP Only (N=398) | DDDRP (N=383)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 0 (0)
Coagulation problem (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Cornary Syndrome/Acute Myocardial Infarction (Cardiac disorders) | 7 (8) | 5 (6) | 5 (5)
Atrial Arrhythmia (Cardiac disorders) | 42 (58) | 50 (71) | 38 (42)
AV conduction disorders (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac death (Cardiac disorders) | 7 (7) | 8 (8) | 8 (8)
General cardiovascular disorders (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
Heart Failure (Cardiac disorders) | 13 (17) | 13 (16) | 13 (16)
Sudden Cardiac Arrest (Cardiac disorders) | 4 (4) | 6 (6) | 3 (3)
Sympthoms of chest pain, angina, palpitation, dyspnea on exertion or cardiopalmo (Cardiac disorders) | 13 (16) | 7 (9) | 8 (8)
Ventricular Tachycardia or Fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 6 (6)
Glucose metabolism disorders (Endocrine disorders) | 3 (3) | 3 (3) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Eye disease (Eye disorders) | 1 (1) | 0 (0) | 3 (3)
Gastrointestinal disorders (Gastrointestinal disorders) | 10 (16) | 5 (6) | 7 (8)
Death for non cardiac reason (General disorders) | 10 (10) | 15 (15) | 8 (8)
Death for unknown causes (General disorders) | 15 (15) | 13 (13) | 25 (25)
Hemorrage (General disorders) | 7 (10) | 6 (7) | 5 (5)
Hypertension (General disorders) | 3 (3) | 4 (4) | 1 (1)
Other general disorders (General disorders) | 20 (24) | 14 (14) | 14 (16)
Syncope (General disorders) | 4 (4) | 4 (4) | 8 (8)
Gallbladdert disorder (Hepatobiliary disorders) | 4 (4) | 0 (0) | 1 (3)
Hepatic disorder (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Infection and infestations (Infections and infestations) | 3 (4) | 4 (4) | 4 (5)
Consequences of drugs administration (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 3 (3)
Lead dislodgement (Injury, poisoning and procedural complications) | 17 (19) | 18 (19) | 15 (15)
Pacemaker/Lead related complications (Injury, poisoning and procedural complications) | 5 (5) | 3 (4) | 4 (4)
Ureteral catheter dysfunction or dislodgement (Injury, poisoning and procedural complications) | 1 (10) | 0 (0) | 0 (0)
Enteroscopy, colonoscopy or video capsule endoscopy procedure (Investigations) | 2 (3) | 0 (0) | 0 (0)
Muscoloskeletal disease (Musculoskeletal and connective tissue disorders) | 23 (33) | 5 (5) | 10 (11)
Neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (11) | 7 (7) | 4 (4)
Prostate disorder (Renal and urinary disorders) | 3 (3) | 2 (2) | 0 (0)
Renal or urinary disease (Renal and urinary disorders) | 4 (4) | 7 (9) | 3 (4)
Acute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 1 (1) | 1 (1)
Cronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 1 (2)
Other respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8) | 8 (8)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 7 (10) | 3 (3)
Symptoms of dyspnea, shortness of breath, fatigue, cough and or tachypnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (7) | 4 (4)
Ablation (Surgical and medical procedures) | 2 (2) | 2 (2) | 3 (3)
Coronary Artery Bypass Graft (Surgical and medical procedures) | 3 (3) | 1 (1) | 0 (0)
Other cardiac surgical interventions (Surgical and medical procedures) | 2 (3) | 3 (3) | 4 (4)
Other surgical interventions (Surgical and medical procedures) | 9 (11) | 21 (22) | 16 (16)
Pacemaker replacement, explant or repositioning (Surgical and medical procedures) | 17 (17) | 7 (7) | 17 (17)
Stent implantation/Angiography (Surgical and medical procedures) | 6 (6) | 3 (3) | 5 (5)
Aneurysm (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Coronary Artery Disease (Vascular disorders) | 2 (2) | 1 (1) | 2 (2)
Other cerebrovascular disorders (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Other vascular disorders (Vascular disorders) | 0 (0) | 3 (4) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Vascular disorders) | 4 (4) | 3 (3) | 2 (2)
Transient Ischemic Attack (Vascular disorders) | 4 (4) | 4 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No